CLINICAL TRIAL: NCT00219193
Title: An Eight Week, Multicenter Study to Evaluate Efficacy and Safety of the Triple Combo of Aliskiren /Valsartan/HCTZ (300/320/25 mg), Compared to the Double Combos of Aliskiren/HCTZ (300/25 mg) or Valsartan/HCTZ (320/25 mg) in Patients With Essential Hypertension Not Adequately Responsive to HCTZ 25 mg
Brief Title: A Clinical Study to Evaluate the Safety and Efficacy of the Combination of Aliskiren and Valsartan in Hypertensive Non Responders Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPP100A2331
Record Dates: First submitted 2005-09-12; First posted 2005-09-22 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Hypertension
Keywords: Hypertension, aliskiren, blood pressure, valsartan, HCTZ
MeSH Terms: conditions — Hypertension | interventions — aliskiren

INTERVENTIONS:
Drug: aliskiren

SUMMARY:
To evaluate the blood pressure lowering effect and safety of the triple combination aliskiren / valsartan / HCTZ (300/320/25 mg) in patients with essential hypertension not adequately responsive to HCTZ 25 mg

ELIGIBILITY:
Inclusion Criteria

* Patients with essential hypertension
* Patients who are eligible and able to participate in the study

Exclusion Criteria

* Severe hypertension
* History or evidence of a secondary form of hypertension

Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 641 (Actual)
Dates: Start 2005-10; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in diastolic blood pressure after 8 weeks

SECONDARY OUTCOMES:
Change from baseline in systolic and diastolic blood pressure after 4 weeks and 8 weeks
Change from baseline in standing blood pressure after 4 weeks and 8 weeks
Achieve blood pressure control target of < 140/90 mmHg after 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States
- Investigative Centers, Germany

REFERENCES:
- [Result] Geiger H, Barranco E, Gorostidi M, Taylor A, Zhang X, Xiang Z, Zhang J. Combination therapy with various combinations of aliskiren, valsartan, and hydrochlorothiazide in hypertensive patients not adequately responsive to hydrochlorothiazide alone. J Clin Hypertens (Greenwich). 2009 Jun;11(6):324-32. doi: 10.1111/j.1751-7176.2009.00114.x. PMID 19527323